CLINICAL TRIAL: NCT03699475
Title: A Randomized Phase II/III Study of αβ T Cell-Depleted, Related, Haploidentical Hematopoietic Stem Cell Transplant (Haplo-HSCT) Plus Rivogenlecleucel vs. Haplo-HSCT Plus Post-Transplant Cyclophosphamide (PTCy) in Patients With AML or MDS
Brief Title: Study of Haplo-HSCT + Rivogenlecleucel vs Haplo-HSCT + Post Transplant Cyclophosphamide in Patients With AML or MDS
Acronym: THRIVE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding, portfolio re-prioritization
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BPX501-301A
Expanded Access: NCT03639844 (No longer available)
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — AP 1903 reagent; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- single-arm Phase II: 3 x 10E6 BPX-501 cell/kg (Experimental): Determining the safety of maximum allowable Dose for BPX-501 starting at 3 x 10E6 cells/kg
  Rimiducid will be administered to inactivate rivogenlecleucel in the event of GVHD not responsive to standard of care treatment
  Interventions: Biological: rivogenlecleucel; Drug: rimiducid; Procedure: haplo-HSCT
- phase 3 Arm A: Dose Determined in phase 2 group (never completed) (Experimental): αβ T cell and CD19+ B cell-depleted, related haploidentical hematopoietic stem cell transplantation (haplo-HSCT) plus rivogenlecleucel
  Interventions: Biological: rivogenlecleucel; Drug: rimiducid; Procedure: haplo-HSCT
- phase 3 Arm B: dose determined in the phase 2 group (never completed) (Active Comparator): haplo-HSCT followed by post-transplant cyclophosphamide (PTCy) in patients with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS)
  Interventions: Drug: Cyclophosphamide; Procedure: haplo-HSCT

INTERVENTIONS:
Biological: rivogenlecleucel — Biological: T cells transduced with caspase 9 safety switch
  Other Names: BPX-501 T cells
  Arms: phase 3 Arm A: Dose Determined in phase 2 group (never completed); single-arm Phase II: 3 x 10E6 BPX-501 cell/kg
Drug: rimiducid — administered to inactivate rivogenlecleucel in the event of GVHD
  Other Names: AP1903
  Arms: phase 3 Arm A: Dose Determined in phase 2 group (never completed); single-arm Phase II: 3 x 10E6 BPX-501 cell/kg
Drug: Cyclophosphamide — GVHD prophylaxis
  Other Names: Cytoxan
  Arms: phase 3 Arm B: dose determined in the phase 2 group (never completed)
Procedure: haplo-HSCT — treatment for disease

SUMMARY:
This study compares the safety and effectiveness of giving rivogenlecleucel (BPX-501 T cells) to patients with AML or MDS post haploidentical hematopoietic stem cell transplant compared to post-transplant cyclophosphamide.

DETAILED DESCRIPTION:
In the Phase 2 portion, participants will undergo αβ T cell and CD19+ B cell depleted haploidentical HSCT followed by an infusion of a fixed dose of rivogenlecleucel (BPX-501 T cells) per kg. These participants will be evaluated for prespecified dose limiting toxicities (DLTs) for a 100-day dose limiting toxicity window.

Following completion of the Phase 2 portion, participants will be enrolled and randomized to one of two treatment arms in the Phase 3 portion.

* Arm A:αβ T-cell and CD19+ B-cell-depleted haplo-HSCT plus treatment with rivogenlecleucel
* Arm B: haplo-HSCT plus post transplant cyclophosphamide

Pediatric patients ages 12-17 will also be included in US only.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent

Meeting institutional criteria to undergo allogenic HSCT

Age 18-70 y/o (12-70 y/o in US only)

Patients with AML or MDS as defined below:

AML Patients Patients with intermediate to adverse AML as defined by ELN (Dohner, 2017).

* AML in first complete remission (CR1) with high-risk features defined as > 1 cycle of induction therapy required to achieve remission OR preceding MDS or myeloproliferative disease
* AML in CR1 with intermediate-risk features
* AML in second or subsequent complete response
* AML with myelodysplasia-related changes (AML-MRC)
* Therapy related AML in first or subsequent complete remission
* De novo AML in second or subsequent complete remission

MDS Patients

* High or very-high risk MDS by IPSS-R classification
* Intermediate risk or higher MDS patients who failed a hypomethylating agent

Lack of suitable conventional donor (i.e. HLA 10/10 related or unrelated donor)

At least a 5/10 genotypic identical haplotype match

The donor and recipient must be identical, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-C, HLA-DRB1, and HLA-DQB1

Patients with adequate organ function

Eastern Cooperative Oncology Group (ECOG) performance status: 0-2

Exclusion Criteria:

* HLA 10/10 allele matched (HLA-A,-B,-C,-DRBl, and DQB1) related donor or unrelated donor
* Autologous hematopoietic stem cell transplant ≤ 3 months before enrollment
* Prior allogeneic transplantation
* Active CNS involvement by malignant cells (less than 2 months from the conditioning)
* Current uncontrolled clinically active bacterial, viral or fungal infection
* Positive HIV serology or viral RNA
* Pregnancy (positive serum or urine βHCG test) or breast-feeding
* Fertile men or women unwilling to use effective forms of birth control or abstinence for a year after transplantation
* Radiographic, histologic, or known history of cirrhosis
* Overlapping MDS and myeloproliferative neoplasms (MPN) disease
* Patients with acute promyelocytic leukemia (APL)
* Known hypersensitivity to dimethyl sulfoxide (DMSO)

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - TriStar Bone Marrow Transplant, LLC, Nashville, Tennessee
  - Methodist Healthcare System of San Antonio Clinical Trials Office, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II, Cohort 1 (Only Study Arm That the Only Participant Enrolled Into): αβ T-cell and CD19+ B-cell-depleted haploidentical stem cell transplantation plus rivogenlecleucel (BPX-501) dose: 3x 10^6 cells/kg
  Rimiducid only to be administered to inactivate rivogenlecleucel in the event of GVHD not responsive to standard of care treatment; (study terminated after enrollment of the first patient total study participant number is 1)
  ---------------------- rivogenlecleucel: Biological: T cells transduced with caspase 9 safety switch
  rimiducid: administered to inactivate rivogenlecleucel in the event of GVHD
  haplo-HSCT: treatment for disease
Period: Overall Study
Arm/Group | Phase II, Cohort 1 (Only Study Arm That the Only Participant Enrolled Into)
Started | 1 (Only a single patient was enrolled to this study which was to the phase 2: Cohort 1 and then the study was terminated early by the Sponsor and no other participants were enrolled in this study in any other group. Therefore, total study participant number is 1.)
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: only 1 patient was enrolled in this study
Groups:
- Phase II, Cohort 1: αβ T-cell and CD19+ B-cell-depleted haploidentical stem cell transplantation plus rivogenlecleucel
  Rimiducid will be administered to inactivate rivogenlecleucel in the event of GVHD not responsive to standard of care treatment
  rivogenlecleucel: Biological: T cells transduced with caspase 9 safety switch
  rimiducid: administered to inactivate rivogenlecleucel in the event of GVHD
  haplo-HSCT: treatment for disease
Arm/Group | Phase II, Cohort 1
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 28 [28 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
history of AML in the second or subsequent complete remission [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing 3 or More Dose Limiting Toxicities [Phase 2] Within a 100-day DLT Window After Receiving BPX-501
Description: If any of the following adverse events that occur within the DLT window they will be considered a DLT:
  * Grade III or IV acute GVHD attributable to rivogenlecleucel and non-responsive to > 1 dose of rimiducid treatment (plus standard doses (at least 1 mg/kg) of methylprednisone or dose equivalent of other corticosteroids, and/or calcineurin inhibitor) within 14 days
  * Grade 3-4 neurologic events attributable to rivogenlecleucel
  * Death due to any cause other than underlying disease
  * Any CTCAE Grade 3-5 adverse events related to rivogenlecleucel (including allergic reactions, infusion reactions, and any other related adverse reactions whether expected or unexpected). in case 3 or more DLTs are observed with 3 x 10E6 dose, another cohort would have been enrolled to receive the 1 x 10E6 cell dose (never happened as study terminated early)
Time Frame: 100 days
Population: Study terminated early after graft failure of the first participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II, Cohort 1
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: from enrolment to 43 days after receiving BPX-501 (subject passed away at this point, study had only enrolled 1 patient)
Description: All AEs were reported. CTCAE version 5.0 was used for grading.
Arm/Group | Phase II, Cohort 1
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II, Cohort 1 (N=1)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1)
Viral sepsis (Infections and infestations) | 1 (1)
Brain hypoxia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II, Cohort 1 (N=1)
Cellulitis (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT03699475/Prot_SAP_001.pdf